CLINICAL TRIAL: NCT01046123
Title: A Phase II Study of Whole Brain Radiotherapy With Simultaneous Integrated Boost Using Volumetric Modulated Arc Therapy for One to Ten Brain Metastases
Brief Title: Volumetric Modulated Arc Therapy (VMAT) for Brain Metastases
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: British Columbia Cancer Agency (Other)
Responsible Party: Principal Investigator, Alan Nichol, Radiation Oncologist, British Columbia Cancer Agency
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WHAM!
Record Dates: First submitted 2010-01-07; First posted 2010-01-11 (Estimated); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Brain Metastases
MeSH Terms: conditions — Brain Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Whole brain radiotherapy (Experimental): whole brain radiotherapy (WBRT) and a simultaneous integrated boost (SIB) using volumetric modulated arc therapy
  Interventions: Radiation: whole brain radiotherapy (WBRT) and a simultaneous integrated boost (SIB) using volumetric modulated arc therapy

INTERVENTIONS:
Radiation: whole brain radiotherapy (WBRT) and a simultaneous integrated boost (SIB) using volumetric modulated arc therapy — Patients will be treated with WBRT/SIB using VMAT, delivering a total of 20 Gy in 5 fractions to the whole brain and 50Gy in 5 fractions to the brain metastases, delivered once daily on working days.

SUMMARY:
Radiotherapy to the whole brain is standard treatment for cancer that has spread to the brain (brain metastases) as it treats both the metastases that can be seen on scans and the brain metastases that are too small to be seen on scans.

This study will use a novel radiotherapy technique, called volumetric modulated arc therapy (VMAT), to treat patients with brain metastases. This technique allows delivery of both a standard radiation dose to the whole brain as well as a higher radiation dose to the brain metastases at the same time.

The study will assess the effectiveness of using VMAT in treating brain metastases, and examine its potential side-effects.

DETAILED DESCRIPTION:
This is a Phase II prospective clinical trial. Following registration, patients will be required to undertake a baseline questionnaire assessment of daily living activities using the Modified Barthel's index, as well as cognitive assessment using MMSE.

Patients will undergo MRI scan of the brain for radiotherapy planning purposes. During radiotherapy planning and for each of the five radiotherapy fractions, patients will be immobilised in a custom fitted stereotactic mask system, to minimise head movement. During treatment, patients will have daily online setup corrections to ensure treatment accuracy.

Patients will be treated with WBRT/SIB using VMAT, delivering a total of 20 Gy in 5 fractions to the whole brain and 50Gy in 5 fractions to the brain metastases, delivered once daily on working days. Anti-nausea and anti-inflammatory medication will be prescribed to minimise acute toxicity.

Following therapy completion, patients will be seen every 3 months for the 1st year, then every 6 months thereafter. At each clinic visit, clinicians or study investigators will monitor for toxicity from therapy, document neurologic symptoms and signs and performance status as well as Modified Barthel's index and cognitive assessment.

Patients will have contrast-enhanced MRI brain at 3 months and 1 year, and contrast-enhanced CT brain at 6 months and 9 months in the first year and every 6 months after the first year. Serum creatinine levels will be done prior to each scan to ensure safety of intravenous contrast administration.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18
* pathologically confirmed solid malignancy diagnosed within the past 5 years (if the original pathological cancer diagnosis is more than 5 years earlier, a biopsy to confirm metastatic relapse within the past 5 years is required)
* 1-10 brain metastases
* Maximum diameter of largest metastasis ≤ 3 cm
* KPS ≥ 70
* Patient is neurologically stable with or without corticosteroids
* Extracranial disease well-controlled (6-month estimated median life expectancy).
* Available for regular clinical and imaging follow up
* Prior craniotomy permitted

Exclusion Criteria:

* Require craniotomy to relieve mass effect
* Previous cranial radiotherapy
* Metastatic germinoma, small cell carcinoma, multiple myeloma, lymphoma or leukaemia.
* Chemotherapy administered within one week before radiotherapy or planned within one week after radiotherapy.
* Metastases within 0.7 cm of the optic chiasm, brainstem or optic nerves
* Brainstem metastases
* Systemic lupus erythematosis, scleroderma, or other connective tissue disorders not in remission
* Multiple sclerosis
* Glomerular Filtration Rate < 60 ml/minute
* Non-small cell lung cancer with liver metastases
* Bilirubin > upper normal limit
* AST or ALT > 2X upper normal limit
* Pregnancy
* Summed volume of all metastasis PTVs > 50 cm3

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2010-01; Primary Completion 2013-06 (Actual); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
3 month treatment response of metastases evaluated using contrast-enhanced MRI scan of brain | 3 months post treatment

SECONDARY OUTCOMES:
1-year local control of treated metastases evaluated with contrast-enhanced MRI scan of brain | 1 year post-treatment
1-year brain control of metastases evaluated with contrast-enhanced MRI scan of brain | 1 year post-treatment
Median survival | No time frame
Both acute neurological toxicity (within 3 months of treatment) and late neurological toxicity (beyond 3 months of treatment | 3 months and beyond
Time to decline in activities of daily living evaluated using the Modified Barthel index | No time frame
Time to decline in cognition evaluated with the Mini-mental state examination | No time frame

CONTACTS AND LOCATIONS:
Overall Officials: Alan M Nichol, MD, Principal Investigator — British Columbia Cancer Agency
Locations (1):
- BC Cancer Agency - Vancouver Centre, Vancouver, British Columbia, Canada

REFERENCES:
- [Derived] Chan M, Ferguson D, Ni Mhurchu E, Yuan R, Gondara L, McKenzie M, Olson R, Thiessen B, Lalani N, Ma R, Nichol A. Patients with pretreatment leukoencephalopathy and older patients have more cognitive decline after whole brain radiotherapy. Radiat Oncol. 2020 Nov 25;15(1):271. doi: 10.1186/s13014-020-01717-x. PMID 33239056
- [Derived] Nichol A, Ma R, Hsu F, Gondara L, Carolan H, Olson R, Schellenberg D, Germain F, Cheung A, Peacock M, Bergman A, Vollans E, Vellani R, McKenzie M. Volumetric Radiosurgery for 1 to 10 Brain Metastases: A Multicenter, Single-Arm, Phase 2 Study. Int J Radiat Oncol Biol Phys. 2016 Feb 1;94(2):312-21. doi: 10.1016/j.ijrobp.2015.10.017. Epub 2015 Oct 22. PMID 26678660